CLINICAL TRIAL: NCT04077606
Title: Gingival Inflammatory Response, Bacterial Adhesion And Patient Satisfaction Of Ceramo-Metallic Vs Zirconia Crowns (Randomized Clinical Study)
Brief Title: Gingival Inflammatory Response,Bacterial Adhesion and Patient Satisfaction of Ceramo-metallic vs Zirconia Crowns
Acronym: CairoU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nashwa Yehia Abd El Badee Hefnawy, Nashwa hefnawy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoUniversity
Record Dates: First submitted 2019-08-19; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Gingival Inflammation; Oral Bacterial Infection
Keywords: interleukin 1 beta, bacterial adhesion,monolithic zirconia
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind (trial participants and outcome assessors). Each participant included in this study will be blinded (without knowing type of intervention received).
  Blinded assessors :blinding to the laboratory assessors is done by not involving them in sequence generation or allocation concealment or treatment options.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceramo-metallic crown (Active Comparator): ceramo-metallic crown preparation
  Interventions: Other: ceramo-metallic crown prepartion; Other: full anatomical monolithic zirconia crown
- monolithic zirconia crown (Active Comparator): monolithic zirconia crown preparation
  Interventions: Other: ceramo-metallic crown prepartion; Other: full anatomical monolithic zirconia crown

INTERVENTIONS:
Other: ceramo-metallic crown prepartion — tooth will be prepared to receive ceramo-metallic crowns
  Other Names: feldspathic porcelain fused to metal
Other: full anatomical monolithic zirconia crown — tooth will be prepared to receive monolithic zirconia crowns
  Other Names: katana zirconia, Kuraray Noritake , Japan

SUMMARY:
Ceramo metallic restoration has proved high success rate over past years as considered to be the gold standard while Monolithic zirconia as fixed dental prostheses have gained attention because of their good fracture strength, low wear of the enamel antagonist and pleasant color .Material composition will affect gingival health and biofilm formation which initiate caries and periodontal diseases.

DETAILED DESCRIPTION:
For years, the ceramo-metal restoration has been the gold standard in crown and bridge procedures .They have been used for many years and studied extensively. Studies have demonstrated a 94% success rate over a 10-year period and good long-term clinical reliability. Although chipping of veneering porcelain is a possible complication, fracture of the metal framework is uncommon . They require sufficient tooth reduction to allow space for at least 0.3 mm of metal coping and 0.7 mm of veneering porcelain, and a minimum facial reduction of 1.2 mm according to Hobo and Shillingburg. When comparing ceramo-metallic crowns to zirconia crowns, several points are noteworthy. Laboratory testing has determined that the fracture strength of a ceramo-metallic crown using 1.5 mm reduction is similar to zirconia crowns with only 1 mm of reduction5. Some manufacturers have even suggested a 0.6 mm minimum reduction for posterior zircona crowns. Which has led some dentists to prescribe all-zirconia restorations to preserve tooth structure6 Zirconia became popular in dentistry because of the material's excellent mechanical properties which include high strength, fracture toughness and biocompatibility.New monolithic CAD/CAM restorative materials are designed to improve the optical and mechanical properties of the avoid veneering failure .To increase translucency and aesthetics of full-contour zirconia ,some modifications ,such as sintering temperature ,fabrication processes and addition of colouring liquids have been applied. These modifications may affect the mechanical and autocatalytic surface-transformation ((low-temperature degradation (LTD)) properties of zirconia.) The primary etiologic factor of gingival inflammation is a plaque, and by inadequate crown shape its accumulation can be facilitated . A single crown can cause inflammation of the periodontal tissue, if the hygienic principles have not been observed during its production. If the finish line of the artificial crown disrupts the biologic width and is placed in the connective tissue attachment area, the inflammation may occur. Even with increased hygiene, the gingival inflammation can occur, if the crown preparation margin is located deeply subgingivally Taking care of the periodontal tissue health the precision of the preparation margin, tightness of proximal contacts, conformity of the tooth crown anatomic shape, occlusal morphology and surface smoothness must be checked . The contact of the crown and the tooth must be tight and uniform .

While choosing material for crown production it must be taken into account that the bacterial adhesive capacity of the prosthetic material is affected by the surface roughness .asperities, free energy of the surface and composition of materials (it is the lowest for ceramic, but the highest for acrylates).Early-colonizing bacteria play a pivotal role for the subsequent adhesion of cariogenic microorganisms such as Streptococcus mutans and periodontal pathogens such as Tannerella forsythensis, Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans, which may induce gingival and periodontal inflammation Periodontal diagnosis generally requires measurement of periodontal tissue destruction (e.g., probing pocket depth [PPD] and clinical attachment level [CAL]) and gingival inflammation (e.g., bleeding on probing [BOP] and gingival index [GI]). Although the techniques used are straightforward and noninvasive. These parameters are static and thus reflect disease history and not present disease activity .Therefore, it is necessary to develop diagnostic tests that can identify active periodontal sites, predict future disease progression, and assess response to periodontal treatment. Periodontopathic bacteria increase the risk of periodontitis, and immune responses against bacterial products and subsequent secretion of proinflammatory cytokines are crucial in periodontal tissue destruction .Interleukin-1β (IL-1β) is an important mediator of inflammatory response and is involved in cell proliferation, differentiation, and apoptosis, and in the pathophysiology of periodontitis.

ELIGIBILITY:
inclusion criteria

* Patient age range from 20-50 to be able to read and write in order to sign the informed consent document.
* Patients physically and psychologically able to tolerate conventional restorative procedures.
* Patients with no active periodontal and or pulpal diseases, having teeth with good restorations.
* Patients with root canal treated teeth requiring full coverage restorations.
* Patients indicated for full coverage (e.g. moderate to severe discoloration, coronal fracture).
* Patients didn't take antibiotics or anti-inflammatory in the past three months.
* Surfaces with an adjacent probing pocket depth exceeding 3mm were not included
* Patients willing to return for follow-up examinations and assessments.

Exclusion criteria:

* Patients in the growth stage with partially erupted teeth.
* Patient with poor oral hygiene.
* Patients with psychiatric problems or unrealistic expectations
* Patient with no opposite occluding dentition in the area intended for restoration.
* Patient suffering from Para functional habits.
* Patient with diabetes mellitus, hypertension and gingivitis or periodontitis which has impact on gingival cervicular fluid level

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Gingival inflammatory response | 12 weeks
  presence and concentration of interleukin 1 -beta

SECONDARY OUTCOMES:
bacterial adhesion | 12 weeks
  colony forming unit

OTHER OUTCOMES:
patient satisfaction | 12 weeks
  patient satisfaction with yes or no

REFERENCES:
- [Background] Griggs JA. Recent advances in materials for all-ceramic restorations. Dent Clin North Am. 2007 Jul;51(3):713-27, viii. doi: 10.1016/j.cden.2007.04.006. PMID 17586152
- [Background] Lekesiz H. Reliability estimation for single-unit ceramic crown restorations. J Dent Res. 2014 Sep;93(9):923-8. doi: 10.1177/0022034514544215. Epub 2014 Jul 21. PMID 25048249
- [Background] Sailer I, Makarov NA, Thoma DS, Zwahlen M, Pjetursson BE. All-ceramic or metal-ceramic tooth-supported fixed dental prostheses (FDPs)? A systematic review of the survival and complication rates. Part I: Single crowns (SCs). Dent Mater. 2015 Jun;31(6):603-23. doi: 10.1016/j.dental.2015.02.011. Epub 2015 Apr 2. PMID 25842099
- [Background] Hobo S, Shillingburg HT Jr. Porcelain fused to metal: tooth preparation and coping design. J Prosthet Dent. 1973 Jul;30(1):28-36. doi: 10.1016/0022-3913(73)90075-9. No abstract available. PMID 4575207
- [Background] Sun T, Zhou S, Lai R, Liu R, Ma S, Zhou Z, Longquan S. Load-bearing capacity and the recommended thickness of dental monolithic zirconia single crowns. J Mech Behav Biomed Mater. 2014 Jul;35:93-101. doi: 10.1016/j.jmbbm.2014.03.014. Epub 2014 Apr 2. PMID 24762856
- [Background] Baladhandayutham B, Lawson NC, Burgess JO. Fracture load of ceramic restorations after fatigue loading. J Prosthet Dent. 2015 Aug;114(2):266-71. doi: 10.1016/j.prosdent.2015.03.006. Epub 2015 May 16. PMID 25985741
- [Background] Piconi C, Maccauro G. Zirconia as a ceramic biomaterial. Biomaterials. 1999 Jan;20(1):1-25. doi: 10.1016/s0142-9612(98)00010-6. PMID 9916767
- [Background] Chen YM, Smales RJ, Yip KH, Sung WJ. Translucency and biaxial flexural strength of four ceramic core materials. Dent Mater. 2008 Nov;24(11):1506-11. doi: 10.1016/j.dental.2008.03.010. Epub 2008 Apr 25. PMID 18440062
- [Background] Beuer F, Schweiger J, Eichberger M, Kappert HF, Gernet W, Edelhoff D. High-strength CAD/CAM-fabricated veneering material sintered to zirconia copings--a new fabrication mode for all-ceramic restorations. Dent Mater. 2009 Jan;25(1):121-8. doi: 10.1016/j.dental.2008.04.019. Epub 2008 Jul 11. PMID 18620748
- [Background] Goldberg PV, Higginbottom FL, Wilson TG. Periodontal considerations in restorative and implant therapy. Periodontol 2000. 2001;25:100-9. doi: 10.1034/j.1600-0757.2001.22250108.x. PMID 11155185
- [Background] Gunay H, Seeger A, Tschernitschek H, Geurtsen W. Placement of the preparation line and periodontal health--a prospective 2-year clinical study. Int J Periodontics Restorative Dent. 2000 Apr;20(2):171-81. PMID 11203559
- [Background] Lang NP, Berglundh T, Heitz-Mayfield LJ, Pjetursson BE, Salvi GE, Sanz M. Consensus statements and recommended clinical procedures regarding implant survival and complications. Int J Oral Maxillofac Implants. 2004;19 Suppl:150-4. No abstract available. PMID 15635955
- [Background] Zenthofer A, Ohlmann B, Rammelsberg P, Bomicke W. Performance of zirconia ceramic cantilever fixed dental prostheses: 3-year results from a prospective, randomized, controlled pilot study. J Prosthet Dent. 2015 Jul;114(1):34-9. doi: 10.1016/j.prosdent.2015.02.006. Epub 2015 Apr 14. PMID 25882973
- [Background] Kato A, Imai K, Ochiai K, Ogata Y. Prevalence and quantitative analysis of Epstein-Barr virus DNA and Porphyromonas gingivalis associated with Japanese chronic periodontitis patients. Clin Oral Investig. 2015 Sep;19(7):1605-10. doi: 10.1007/s00784-014-1387-y. Epub 2014 Dec 18. PMID 25515271
- [Background] Reddy MS. The use of periodontal probes and radiographs in clinical trials of diagnostic tests. Ann Periodontol. 1997 Mar;2(1):113-22. doi: 10.1902/annals.1997.2.1.113. PMID 9151548